CLINICAL TRIAL: NCT02933281
Title: MTBVAC Phase 1b/2a Randomized, Double-blind, Active-controlled,Safety, Immunogenicity, and Dose-escalation Study in Adults With and Without Latent Tuberculosis Infection in South Africa
Brief Title: MTBVAC Study in Adults With and Without Latent Tuberculosis Infection in South Africa
Acronym: A-050
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Biofabri, S.L (Industry); Universidad de Zaragoza (Other); South African Tuberculosis Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A-050
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: MTBVAC 5 x 10^3 CFU (Experimental): Quantiferon (QFT) negative, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 2: MTBVAC 5 x 10^4 CFU (Experimental): QFT Negative, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 3: MTBVAC 5 x 10^5 CFU (Experimental): QFT Negative, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 4: MTBVAC 5 x 10^6 CFU (Experimental): QFT Negative, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 5: MTBVAC 5 x 10^3 CFU (Experimental): QFT Positive, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 6: MTBVAC 5 x 10^4 CFU (Experimental): QFT Positive, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 7: MTBVAC 5 x 10^5 CFU (Experimental): QFT Positive, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- Cohort 8: MTBVAC 5 x 10^6 CFU (Experimental): QFT Positive, 1 dose on Day 0
  Interventions: Biological: MTBVAC
- BCG 5 x 10^5 CFU (Active Comparator): Both QFT positive and negative, 1 dose on Day 0
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: MTBVAC — Escalating dose levels (5 x 10^3 CFU, 5 x 10^4 CFU, 5 x 10^5 CFU, and 5 x 10^6 CFU
  Arms: Cohort 1: MTBVAC 5 x 10^3 CFU; Cohort 2: MTBVAC 5 x 10^4 CFU; Cohort 3: MTBVAC 5 x 10^5 CFU; Cohort 4: MTBVAC 5 x 10^6 CFU; Cohort 5: MTBVAC 5 x 10^3 CFU; Cohort 6: MTBVAC 5 x 10^4 CFU; Cohort 7: MTBVAC 5 x 10^5 CFU; Cohort 8: MTBVAC 5 x 10^6 CFU
Biological: BCG — BCG 5 x 10^5 CFU
  Other Names: BCG 5 x 10^5 CFU
  Arms: BCG 5 x 10^5 CFU

SUMMARY:
MTBVAC at four dose levels: 5 x 10^3 CFU, 5 x 10^4 CFU, 5 x 10^5 CFU, and 5 x 10^6 CFU. The active control is BCG (5 x 10^5 CFU). Participants will receive a single dose of MTBVAC or BCG revaccination administered intradermally on Study Day 0.

DETAILED DESCRIPTION:
This is a Phase 1b/2a, double-blind, randomized, BCG-controlled, dose-escalation safety and immunogenicity study in 144 healthy adults with and without LTBI. All participants will have received previous BCG vaccination in infancy. The investigational product is MTBVAC at four dose levels: 5 x 10^3 CFU, 5 x 10^4 CFU, 5 x 10^5 CFU, and 5 x 10^6 CFU. The active control is BCG (5 x 10^5 CFU).

Participants meeting the inclusion/exclusion criteria will be randomized within a study cohort to receive a single dose of MTBVAC or BCG revaccination administered intradermally on Study Day 0. The study will be conducted at one site in South Africa. Participants will be enrolled into one of eight cohorts and followed for safety and immunogenicity endpoints through Study Day 365. The estimated time to complete enrolment is approximately 12 months.

Cohorts 1-8 will include 72 QFT-negative (Cohorts 1-4) and 72 QFT-positive (Cohorts 5-8) participants. Participants will be randomized within each cohort, to receive either MTBVAC (N=96) or BCG (N=48). The cohorts will be enrolled as described in the protocol, as long as no pausing/stopping rules are triggered

ELIGIBILITY:
Inclusion Criteria

1. Has completed the written informed consent process.
2. Is male or female aged 18 through 50 years on Study Day 0.
3. Agrees to stay in contact with the clinical trial site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study.
4. For female participants: agrees to avoid pregnancy from 21 days prior to Study Day 0 and for the full duration of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, or intrauterine device (IUD).
5. For male participants: agrees to use barrier contraception with his partner for at least 2 weeks after dosing with MTBVAC or BCG.
6. Has general good health, confirmed by medical history and physical examination.
7. Had BCG vaccination, documented through medical history or presence of scar.
8. Has not shared enclosed living or work space with someone diagnosed with TB during the 3 months prior to Study Day 0.
9. [Cohorts 1-4] Does not have LTBI, determined by a negative QFT test at screening or [Cohorts 5-8] Has LTBI, determined by a positive QFT test at screening.

Exclusion Criteria

1. Acute illness on Study Day 0.
2. Axillary temperature >or= 37.5C on Study Day 0.
3. Abnormal laboratory values from most recent blood collection prior to Study Day 0 randomization that are equivalent to Grade 2 or more toxicity, per the protocol toxicity table, or if deemed clinically significant.
4. Severe anemia, defined as <10 g/dL hemoglobin or hematocrit <30%.
5. Screening thyroid stimulating hormone (TSH) >upper limit of normal per local laboratory range.
6. Suspicion or evidence (including but not limited to sputum Xpert MTB/RIF positive) of active TB disease at any site. An attempt must be made to obtain sputum from each participant; persons who are sputum unproductive will be assumed to be Xpert MTB/RIF negative.
7. History of treatment for TB disease.
8. History of autoimmune disease or immunosuppression.
9. Used immunosuppressive medication within 42 days before Study Day 0 (inhaled and topical corticosteroids are permitted).
10. Received immunoglobulin or blood products within 42 days before Study Day 0.
11. Received any investigational drug or investigational vaccine within 182 days before Study Day 0, or planned participation in any other investigational study during the study period.
12. Received investigational vaccine against TB at any time prior to Study Day 0.
13. Planned administration/administration of a licensed vaccine in the period starting 28 days before and ending 28 days after dosing with investigational product.
14. History or laboratory evidence of any past, present, or future possible immunodeficiency state including but not limited to any laboratory indication of HIV-1 infection.
15. History of allergic disease or reactions, including eczema, likely to be exacerbated by any component of the investigational product.
16. Previous medical history that may compromise the safety of the participant in the study, including but not limited to: impairment of pulmonary function from TB infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; uncontrolled epilepsy or infantile spasms; or diabetes mellitus.
17. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine, including axillary lymphadenopathy.
18. Female participants: currently pregnant or lactating/nursing; or positive urine pregnancy test during screening or pre-vaccination on Study Day 0.
19. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, could endanger the participant or make it unlikely that the participant will comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity of MTBVAC at escalating dose levels compared to BCG vaccine by assessing number of participants with AEs and SAEs | Study Days 0 to Day 365
  Collection of systemic solicited and unsolicited adverse events; solicited and unsolicited injection site reactions; and serious adverse reactions.

SECONDARY OUTCOMES:
Difference in T cell response between MTBVAC dose levels across all post-immunization time points measured by percentage of MTBVAC-specific CD4 and CD8 T cells that produce any or a combination of relevant cytokines in ICS assay | Study Days 0, 28, 56, 182, and 365
  12 hour whole blood (WB) intracellular cytokine staining (ICS) assay
Qualitative and quantitative results from QuantiFERON® TB (QFT) test summarized using participant count (percentage) summaries conversion and reversion rates in participants receiving escalating dose levels of MTBVAC | Screening and Study Day 365 (all cohorts); and Study Days 28, 56, 84, and 182 (Cohorts 1-4)
  QFT Gold Plus assay
Qualitative and quantitative results from QFT test using percentage conversion and reversion rates of participants receiving escalating dose levels of MTBVAC compared to BCG dose levels of MTBVAC in comparison to BCG measured by QFT Gold Plus assay | Screening and Study Day 365 (all cohorts); and Study Days 28, 56, 84, and 182 (Cohorts 1-4)
  QFT Gold Plus assay

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Luabeya, MD, Principal Investigator — SATVI
Locations (1):
- SATVI: Worcester, Worcester, South Africa

IPD SHARING:
Plan to Share IPD: No